CLINICAL TRIAL: NCT02692300
Title: Protocol for the Electroencephalography Guidance of Anesthesia to Alleviate Geriatric Syndromes (ENGAGES-CANADA) Study: a Pragmatic, Randomized Clinical Trial
Brief Title: EEG Guidance of Anesthesia (ENGAGES-CANADA)
Acronym: ENGAGES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Queen's University (Other); University of Washington (Other); University of Toronto (Other); Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HS18290
Record Dates: First submitted 2016-02-02; First posted 2016-02-26 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Post-operative Delirium
Keywords: anesthesia; delirium; surgery; electroencephalography; burst suppression; PTSD; anxiety; depression; falls
MeSH Terms: conditions — Emergence Delirium; Delirium; Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Anesthesia practitioner is not blinded to intervention. Subject is blinded and primary outcome assessor is blinded to intervention.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Patients will undergo standard anesthesia and will be blinded to EEG-based data, as per standard of care in this patient population.
- EEG-Guided Group (Experimental): Practitioners will follow the EEG-Guided protocol to limit the incidence of EEG burst suppression by decreasing administration of anesthesia. The EEG-guided protocol is suggestive rather than prescriptive, and practitioners will exercise judgment depending on the clinical situation.
  Interventions: Procedure: EEG-Guided Group

INTERVENTIONS:
Procedure: EEG-Guided Group — Device: Bispectral Index (BIS) processed electroencephalogram or MASIMO or NeuroSENSE
  Arms: EEG-Guided Group

SUMMARY:
This study examines the potential link between deep levels of anesthesia and delirium.

DETAILED DESCRIPTION:
ENGAGES CANADA is a parallel study to the ENGAGES study which has been published in JAMA, DOI:10.1001/jama.2019.5161. Due to the difference in practice models and types of anesthesia principles, ENGAGES CANADA is an important study. Delirium is a relatively common postoperative complication in the geriatric population, affecting 20% to 70% of surgical patients over the age of 60. Delirium manifests as confusion, inattention and the inability to think logically, and may affect the patient's postoperative healing and rehabilitation. It is associated with persistent cognitive decline, longer hospital stay, increased incidence of injurious falls, and increased mortality. Patients undergoing major cardiac surgery are at a significant risk of postoperative delirium. To date, there is no proven method to prevent postoperative delirium in this patient population and often delirious events remain unrecognized. Randomized controlled studies in diverse surgical patient populations suggest that intraoperative electroencephalography (EEG) guidance during general anesthesia may decrease postoperative delirium and adverse postoperative outcomes. Patients who experience postoperative delirium report persistently decreased quality of life and it is a risk factor for incident psychiatric disorders and psychotropic medication use. One potential key mechanism in the relationship between delirium and incident psychiatric illness may be the experience of dissociation (disturbed awareness, impaired memory, or altered perceptions) in the perioperative period in those who are delirious. The co-occurrence of psychiatric illness and delirium can put older adults at greater risk of negative long terms effect such as functional decline. This study will compare the effectiveness of two anesthetic protocols in reducing postoperative delirium and postoperative health-related quality of life in a high risk population.We expect that EEG-guided anesthetic management of patients during their operative procedure will result in improved health-related outcomes, specifically decreased incidence of postoperative delirium and improved postoperative mental and physical health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 60 years or older;
2. Competent to provide informed consent;
3. Undergoing elective cardiac surgery requiring cardiopulmonary bypass.

Exclusion Criteria:

1. Unable to provide informed consent;
2. Preoperative delirium;
3. Unable to participate adequately in delirium screening including those who are blind, deaf, illiterate or not fluent English or French;
4. History of intraoperative awareness

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1225 (Actual)
Dates: Start 2016-12-28 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Incidence of post-operative delirium | 5 days
  Incidence of delirium will be compared between the Control Group and the EEG-Guided Group as measured by the numbers of positive Confusion Assessment Method (CAM) or CAM for intensive care unit (CAM-ICU) scores, coupled with Chart Review.

SECONDARY OUTCOMES:
Incidence of mortality at 30 days and at 1 year | 30 days, 1 year
  Incidence of mortality (%) will be compared between the Control Group and the EEG-Guided Group at 30 days and at 1 year
Length of ICU stay | Time (days) in ICU from Post-Operative Day (POD) 1 to 5 (or through study completion at one year)
  Length of ICU stay (days) will be compared between the Control Group and the EEG-Guided Group.
Length of Hospital stay | Time (days) from admission to discharge from hospital (or through study completion at one year)
  Length of hospital stay (days) will be compared between the Control Group and the EEG-Guided Group.

OTHER OUTCOMES:
Incidence of falls at 30 days and 1 year | 30 days, 1 year
  Number of falls will be recorded by patient interview at 30 days and 1 year, compared between the Control Group and the EEG-Guided Group.
Duration of delirium | 5 days
  Time (days) measured between the first and last positive CAM assessments and compared between the Control Group and the EEG-Guided Group.
Severity of delirium | 5 days
  Severity of delirium will be compared between the Control Group and the EEG-Guided Group. As assessed by the CAM-S severity score
Association between delirium and falls | 30 days and 1 year
  The overall incidence of delirium as assessed by CAM vs the incidence of falls by an adjusted regression model.
Association between delirium and quality of life by PROMIS Global Health | 30 days and 1 year
  The overall incidence of delirium as assessed by CAM vs quality of life as assessed by the PROMIS Global Health measure, by an adjusted regression model.
Predictors and outcomes of perioperative dissociation by PDEQ at 5 days and 30 days postoperatively. | 5 day and 30 days
  A regression model will be used to assess independent predictors of dissociation as assessed by the PDEQ measure, and mental health outcomes associated with perioperative dissociation.
Predictors and outcomes of perioperative distress by PDI at 5 days and 30 days postoperatively | 5 days and 30 days
  A regression model will be used to assess independent predictors of PTSD as assessed by the PDI measure.
Association between depth of anesthesia by EEG monitoring and mortality rate | 1 year
  Depth of anesthesia measured by BIS, Medline, or MASIMO monitors vs mortality rate by an adjusted regression model.
Predictors of Post-Traumatic Stress Disorder (PTSD) using the Post-Traumatic Checklist for DSM-5 (PCL-5). | 30 days and 1 year
  A regression model will be used to assess independent predictors of PTSD as assessed by the PCL-5 measure. This score predicts the risk of PTSD from 0, negligible risk, to 80, extremely high risk of PTSD in patients.
Incidence of major intraoperative and postoperative complications. | Up to 30 days post surgery
  Undesirable intraoperative movement, awareness with recall, complications such as major blood loss and transfusions, stroke, sternal wound infection, sepsis, dialysis, prolonged intubation

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jacobsohn, MBChB FRCPC, Study Director — University of Manitoa; Michael Avidan, MBBCh FCASA, Study Director — Washington University School of Medicine; Tarit Saha, MD FRCPC, Study Director — Queens University; Alain Deschamps, PhD MD FRCPC, Principal Investigator — Université de Montréal; George Djaiani, MD, Study Director — University of Toronto; Renée El-Gabalawy, MA PhD, Study Director — University of Manitoba
Locations (1):
- Montreal Heart Institute, Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deschamps A, Ben Abdallah A, Jacobsohn E, Saha T, Djaiani G, El-Gabalawy R, Overbeek C, Palermo J, Courbe A, Cloutier I, Tanzola R, Kronzer A, Fritz BA, Schmitt EM, Inouye SK, Avidan MS; Canadian Perioperative Anesthesia Clinical Trials Group. Electroencephalography-Guided Anesthesia and Delirium in Older Adults After Cardiac Surgery: The ENGAGES-Canada Randomized Clinical Trial. JAMA. 2024 Jul 9;332(2):112-123. doi: 10.1001/jama.2024.8144. PMID 38857019
- [Derived] Deschamps A, Saha T, El-Gabalawy R, Jacobsohn E, Overbeek C, Palermo J, Robichaud S, Dumont AA, Djaiani G, Carroll J, Kavosh MS, Tanzola R, Schmitt EM, Inouye SK, Oberhaus J, Mickle A, Ben Abdallah A, Avidan MS, Clinical Trials Group CPA. Protocol for the electroencephalography guidance of anesthesia to alleviate geriatric syndromes (ENGAGES-Canada) study: A pragmatic, randomized clinical trial. F1000Res. 2019 Jul 23;8:1165. doi: 10.12688/f1000research.19213.2. eCollection 2019. PMID 31588356